CLINICAL TRIAL: NCT03961204
Title: Evaluating the Long-Term Outcomes and Durability of Effect Following Treatment With Cladribine Tablets for MS: An Exploratory Phase IV Ambispective Study of Patients Who Previously Participated in the CLARITY/CLARITY-EXT and ORACLE MS Clinical Trials (CLASSIC-MS)
Brief Title: Long-Term Outcomes and Durability of Effect Following Treatment With Cladribine Tablets for MS (CLASSIC-MS)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: EMD Serono Research & Development Institute, Inc. (Industry)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Organization: EMD Serono (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MS700568_0026; 2019-000069-19 (EudraCT Number)
Record Dates: First submitted 2019-05-22; First posted 2019-05-23 (Actual); Results first posted 2022-05-05 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Multiple Sclerosis (MS)
Keywords: Multiple Sclerosis; Cladribine; High Disease Activity
MeSH Terms: conditions — Multiple Sclerosis | interventions — Data Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Cohort A (Other): The participants previously enrolled in parent studies CLARITY (NCT00213135), CLARITY-EXT (NCT00641537), ORACLE (NCT00725985) and had received Cladribine tablet and Placebo were invited up to 2 visit for follow-up/data collection.
  Interventions: Other: Data Collection

INTERVENTIONS:
Other: Data Collection — No study treatment was administered as part of this study

SUMMARY:
The objective of this study was to collect data both retrospectively and prospectively in order to evaluate the long-term outcomes, durability of effect, and real-world treatment patterns following treatment with Cladribine Tablets or placebo in participants with multiple sclerosis (MS) who were previously participated in the parent studies (ORACLE MS and CLARITY/CLARITY-EXT).

ELIGIBILITY:
Inclusion Criteria:

* Participants with relapsing remitting multiple sclerosis (RRMS) randomised in CLARITY/CLARITY-EXT clinical trial(s) who have received greater than or equal to (>=) 1 course of in investigational medicinal product (IMP) Cladribine Tablets or placebo
* Participants with their first clinical demyelinating event randomised in ORACLE MS clinical trial who have received >= 1 course of IMP Cladribine Tablets or placebo
* Participants who has sign informed consent which includes compliance with the requirements and restrictions listed in the informed consent form and this protocol

Exclusion Criteria:

* Participants who has any uncontrolled disease state other than MS, that in the Investigator's opinion, constitutes an inappropriate risk or a contraindication for participation in the study or that could interfere with the study objectives, conduct, or evaluation
* For study participants at selected sites where MRI assessment will be conducted following exclusion criteria will apply to MRI assessments only:
* Female study participants who are pregnant
* Participants who are taking Cladribine Tablets as part of another study at the time of the start of this study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 662 (Actual)
Dates: Start 2019-08-15 (Actual); Primary Completion 2021-02-27 (Actual); Study Completion 2021-05-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany
Locations (99):
- United States (7):
  - MS Center of Atlanta, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - University of Maryland, Baltimore - Maryland Center for MS, Baltimore, Maryland
  - Empire Neurology, PC - Empire Neurology PC, Latham, New York
  - Sanford Neuro Health Center - Neurology, Fargo, North Dakota
  - OMRF, Oklahoma City, Oklahoma
  - Rowan University School of Osteopathic Medicine - Department of Medicine, Philadelphia, Pennsylvania
- University of Sydney, Camperdown, Australia
- Barmherzige Brueder Konventspital Linz - Abteilung fuer Neurologie, Linz, Austria
- Belgium (2):
  - Limburgs Universitair Centrum, Hasselt
  - University Hospital of Liege, Seraing
- Bulgaria (5):
  - Military Medical Academy - MHAT - Pleven, Pleven
  - MHAT - Shumen, AD, Shumen
  - MHAT - "National Heart Hospital" EAD - Multiple Clinics, Sofia
  - University Hospital "Saint Naum", Sofia
  - Multiprofile Hospital for Active Treatment - Stara Zagora, Stara Zagora
- Canada (4):
  - Burnaby Hospital Vancouver, Burnaby
  - Clinique Neuro-Outaouais, Gatineau
  - Recherche Sepmus, Inc., Greenfield Park
  - The Ottawa Hospital - General Campus, Ottawa
- Croatia (2):
  - Clinical Hospital Centar Split, Split
  - General Hospital Varazdin, Varaždin
- Czechia (6):
  - Privatni ordinace - neurologie - Nestatni zdravotnicke zarizeni, Hradec Králové
  - Fakultni nemocnice Olomouc - Neurologicka klinika, Olomouc
  - Fakultni nemocnice Ostrava - Dept of Neurology, Ostrava-Poruba
  - Fakultni nemocnice v Motole - Interní klinika 2. LF UK a FN Motol, Prague
  - Vseobecna fakultni nemocnice v Praze - Dept of Neurologicka klinika 1.LF UK a VFN v Praze, Prague
  - Krajska zdravotni, a.s. - Nemocnice Teplice, o.z. - Neurologicke oddeleni, Teplice
- Estonia (2):
  - Astra Team Clinic, Tallinn
  - Tartu University Hospital, Tartu
- Neuro NEO Oy - NEO Research, Turku, Finland
- France (3):
  - Hopital Roger Salengro - CHU Lille - service de neurologie D, Lille
  - CHU de Nîmes - Hôpital Carémeau - Service de Neurologie, Nîmes
  - CHU Rennes - Hopital Pontchaillou - Neurologie - Clinique Neurologique, Rennes
- Georgia (2):
  - Ltd. Pineo Medical Ecosystem, Tbilisi
  - S. Khechinashvili University Clinic, Tbilisi
- Germany (4):
  - Heinrich-Heine-Universitaet Duesseldorf - Klinik fuer Nephrologie, Düsseldorf
  - Diakoniekrankenhaus Henriettenstiftung GgmBH, Hanover
  - Klinik Und Poliklinik Fur Neurologie, Regensburg
  - Universitaetsmedizin Rostock - Klinik und Poliklinik fuer Neurologie, Rostock
- Italy (12):
  - Azienda Ospedaliero Universitaria Consorziale Policlinico di Bari - Neurofisiopatologia, Bari
  - A.O.U. Policlinico V. Emanuele - Presidio Gaspare Rodolico - Clinica Neurologica I, Catania
  - Ospedale Clinicizzato SS. Annunziata - Centro Regionale Sclerosi Multipla, Chieti
  - Azienda Socio Sanitaria Territoriale della Valle Olona (presidio di Gallarate), Gallarate
  - Azienda Ospadaliero Universitaria San Martino - PARENT, Genova
  - Ospedale San Raffaele - U.O. di Neurologia, Milan
  - Azienda Ospedaliera Universitaria "Federico II" - Gastroenterologia Pediatrica, Napoli
  - Azienda Ospedaliero_Universitaria S. Luigi Gonzaga - Centro di Riferimento Regionale Sclerosi Multipla, Orbassano
  - Fondazione Istituto Neurologico Casimiro Mondino - Unità Complessa Malattie Cerebrovascolari/Stroke U, Pavia
  - Azienda Ospedaliera San Camillo Forlanini, Roma
  - Azienda Ospedaliera Universitaria Policlinico Tor Vergata - Dip. Neuroscienze-Centro per la Sclerosi Multipla, Roma
  - Ospedale Sant'Andrea di Roma - MS Center, Rome
- Lebanon (2):
  - American University of Beirut Medical Center, Beirut
  - Bellevue Medical Center, Beirut
- Hospital of Lithuanian University of Health Sciences Kaunas Clinics - Neurology Clinic, Kaunas, Lithuania
- Norway (2):
  - Department of Neurology, Haukeland University, Haukeland
  - St Olavs Hospital - PARENT, Trondheim
- Poland (5):
  - Szpital im. Mikołaja Kopernika - Neurology, Gdansk
  - Uniwersyteckie Centrum Kliniczne - Dept of Neurology, Gdansk
  - Prof. Dr. med. Zbigniew Stelmasiak Specjalistyczny Gabinet Neurologiczny, Lublin
  - Szpital Kliniczny im.Heliodora Swiecickiego Uniwersytetu Medycznego im.K. Marcinkowskiego w Poznaniu - Dept of Neurology, Poznan
  - Instytut Psychiatrii i Neurologii, Warsaw
- Centro Hospitalar de Lisboa Central, E.P.E. - Hospital de Santo António dos Capuchos - Serviço de Neurologia, Lisbon, Portugal
- Romania (3):
  - SC Sana Monitoring SRL., Bucaresti
  - Spitalul Clinic Judetean de Urgenta Targu Mures - Sectia Clinica Neurologie I, Târgu Mureş
  - Spitalul Clinic Judetean de Urgenta "Pius Branzeu" Timisoara - Clinica de Neurologie II, Timișoara
- Russia (18):
  - SAIH "Kemerovo Regional Clinical Hospital" - PARENT, Kemerovo
  - BMI "Kursk Regional Clinical Hospital", Kursk
  - NHI "Central Clinical Hospital #2 of JSC "Russian Railways" n.a. N.A. Semashko, Moscow
  - SBIH of Moscow "City Clinical Hospital # 24" - Branch 1, Moscow
  - SBIH of Moscow region " Moscow Regional Scientific and Research Clinical Institute n.a. M.F. Vladimi, Moscow
  - Medis, Nizhny Novgorod
  - RSHI"State Novosibirsk Regional Clinical Hospital", Novosibirsk
  - SEIHPE "Rostov State Medical University of MoH of RF", Rostov-on-Don
  - LLC " International Clinic MEDEM", Saint Petersburg
  - Pavlov First Saint Petersburg State Medical University - PARENT, Saint Petersburg
  - Saint-Petersburg SU on b.o. City Multifield Hospital #2 - Intensive Pulmonology and Thoracal Surgery, Saint Petersburg
  - SBIH "Leningrad Regional Clinical Hospital", Saint Petersburg
  - SBIH "Samara Regional Clinical Hospital n.a. V.D. Seredavin, Samara
  - SBEI HPE "Saratov State Medical University n.a. V. I. Razumovskiy" of the MoH of the RF, Saratov
  - RSBIH "Smolensk Regional Clinical Hospital", Smolensk
  - Siberian State Medical University, Tomsk
  - Regional Multiple Sclerosis Centre b/o CC ECM "Neftyanik" - Neurology, Tyumen
  - SBHI of Yaroslavl Region "Clinical Hospital # 8" - Cardiology, Yaroslavl
- Serbia (2):
  - Clinical Center of Serbia, Belgrade
  - Clinical Center Nis - Clinic of Neurology, Niš
- South Korea (2):
  - National Cancer Center, Goyang-si
  - Severance Hospital, Yonsei University, Seoul
- Spain (2):
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital Universitario Nuestra Señora de la Candelaria - Servicio de Neurologia, Santa Cruz de Tenerife
- Sahlgrenska Sjukhuset, Gothenburg, Sweden
- (CHUV), Centre Hospitalier Universitaire Vaudois - Departement des Neurosciences Cliniques, Lausanne, Switzerland
- Tunisia (3):
  - Hôpital Fattouma Bourghiba, Monastir
  - Hôpital Habib Bourguiba - Service de Neurologie, Sfax
  - Hopital Militaire de Tunis, Tunis
- Ukraine (2):
  - SI Institute of Neurology, Psychiatry and Narcology of NAMSU - Dept of Neuroinfections and Multiple Sclerosis, Kharkiv
  - Vinnitsa State Medical University - Neurology dept, Vinnytsia
- United Kingdom (2):
  - Nottingham University Hospital - Division of Clinical Neurology, Nottingham
  - Royal Hallamshire Hospital - Dept of Neurology, Sheffield

IPD SHARING:
Plan to Share IPD: Yes
Per company policy, following approval of a new product or a new indication for an approved product in both the EU and the US, EMD Serono will share study protocols, anonymized patient level and study level data and redacted clinical study reports from clinical trials in patients with qualified scientific and medical researchers, upon request, as necessary for conducting legitimate research. Further information on how to request data can be found on our website https://www.emdgroup.com/en/research/our-approach-to-research-and-development/healthcare/clinical-trials/commitment-responsible-data-sharing.html
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Within six months after the approval of a new product or a new indication for an approved product in both the United States and the European Union
Access Criteria: Qualified scientific and medical researchers can request the data. Such requests must be submitted in writing to the company's portal and will be internally reviewed regarding criteria for researchers' qualification and legitimacy of the research proposal.
URL: https://bit.ly/IPD21

REFERENCES:
- [Result] Giovannoni G, Boyko A, Correale J, Edan G, Freedman MS, Montalban X, Rammohan K, Stefoski D, Yamout B, Leist T, Aydemir A, Borsi L, Verdun di Cantogno E. Long-term follow-up of patients with relapsing multiple sclerosis from the CLARITY/CLARITY Extension cohort of CLASSIC-MS: An ambispective study. Mult Scler. 2023 May;29(6):719-730. doi: 10.1177/13524585231161494. Epub 2023 Apr 3. PMID 37012898
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=MS700568_0026
- See also: US Medical Information website, Medical Resources — https://medical.emdserono.com/en_US/home.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 662 subjects were enrolled in this trial at different sites in United States and Europe.
Groups:
- Cohort A: Participants previously enrolled in parent studies CLARITY (NCT00213135), CLARITY-EXT (NCT00641537), ORACLE (NCT00725985) and had received Cladribine tablet and Placebo were invited up to 2 visit for follow-up/data collection.
Period: Overall Study
Arm/Group | Cohort A
Started | 662
Completed | 655
Not Completed | 7
Not completed — Withdrawal by Subject | 2
Not completed — Lost to Follow-up | 3
Not completed — Other | 1
Not completed — Missing | 1

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all participants participating in CLASSIC study [randomized in CLARITY and have received ≥ 1 course of investigational medicinal product (IMP) (Cladribine Tablets or placebo) or participants randomized in the ORACLE study and have received ≥ 1 course of IMP].
Arm/Group | Cohort A
Number analyzed (Participants) | 662
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.3 (10.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 444
  Male | 218
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 8
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 645
  More than one race | 6
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Using Wheelchair or Being Bedridden Assessed by Expanded Disability Status Scale (EDSS) Score 7.0 or Higher
Description: EDSS is a scale based on standardized neurological examination which comprised of optic, brain stem, pyramidal, cerebellar, sensory & cerebral functions, as well as walking ability. EDDS is a scale from 0-10 that evaluates a person with Multiple Sclerosis (MS) disability/neurologic function level where 0=normal and 10=death due to MS. Score of 7.0 is defined as unable to walk beyond approximately 5 meters even with aid, essentially restricted to wheelchair; wheels self in standard wheelchair and transfers alone; up and about in wheelchair some 12 hours a day. Score of 8.0 is defined as Essentially restricted to bed or chair or perambulated in wheelchair, but may be out of bed itself much of the day; retains many self-care functions; generally has effective use of arms.
Time Frame: 3 months prior to study visit 1. Retrospectively from end of parent study (NCT00213135, NCT00641537 and NCT00725985) to study visit 1 (study visit 1 occurred up to 3 months from screening)
Population: FAS included all participants participating in CLASSIC study [randomized in CLARITY and have received ≥ 1 course of investigational medicinal product (IMP) (Cladribine Tablets or placebo) or participants randomized in the ORACLE study and have received ≥ 1 course of IMP]. Number of participants analyzed signifies number of participants who were evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participant
Arm/Group | Cohort A
Number analyzed (Participants) | 636
percentage of participant | 8.2 [6.2 to 10.6]

2. Secondary Outcome: Percentage of Participants With Expanded Disability Status Scale (EDSS) Score 6.0 or Higher
Description: EDSS is a scale based on standardized neurological examination which comprised of optic, brain stem, pyramidal, cerebellar, sensory & cerebral functions, as well as walking ability. EDDS is a scale from 0-10 that evaluates a person with MS disability/neurologic function level where 0= normal and 10= death due to MS. Score of 6.0 is defined as "intermittent or unilateral constant assistance (cane, crutch and brace) required to walk about 100 meters with or without resting".
Time Frame: At study visit 1. Retrospectively after last IMP administration from parent study (NCT00213135, NCT00641537 and NCT00725985) to study visit 1 (study visit 1 occurred up to 3 months from screening)
Population: FAS included all participants participating in CLASSIC study [randomized in CLARITY and have received ≥ 1 course of IMP (Cladribine Tablets or placebo) or participants randomized in the ORACLE study and have received ≥ 1 course of IMP].
Measure: Number (95% Confidence Interval); unit: percentage of participant
Arm/Group | Cohort A
Number analyzed (Participants) | 662
percentage of participant | 13.9 [11.4 to 16.8]

3. Secondary Outcome: Clinical and Demographic Characteristic: Age, Disease Duration
Description: Clinical and demographic characteristics including age and disease duration is reported in the form of long term responders and non-responder. Here long term responder is defined as study participants not requiring disease modifying drug (DMD) 4 years or later following their last dose of IMP in parent study. Non-responder is defined as study participants requiring DMD less than 4 years following their last dose of IMP in parent study.
Time Frame: At study visit 1, occurred up to 3 months from screening (Retrospective analysis of medical record of parent study-NCT00213135, NCT00641537 and NCT00725985)
Population: FAS included all participants participating in CLASSIC study [randomized in CLARITY and have received ≥ 1 course of IMP (Cladribine Tablets or placebo) or participants randomized in the ORACLE study and have received ≥ 1 course of IMP]. Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure and and "Number analyzed" refers to number of participants evaluable for specified categories.
Measure: Mean (Standard Deviation); unit: years
Arm/Group | Cohort A
Number analyzed (Participants) | 627
years
  Long-term responders: Age at study visit 1: number analyzed (Participants) | 378
  Long-term responders: Age at study visit 1 | 50.5 (10.65)
  Non-responders: Age at study visit 1: number analyzed (Participants) | 249
  Non-responders: Age at study visit 1 | 47.1 (9.47)
  Long term responder: Disease duration: number analyzed (Participants) | 330
  Long term responder: Disease duration | 19.82 (9.161)
  Non-responder: Disease duration: number analyzed (Participants) | 226
  Non-responder: Disease duration | 16.82 (8.321)

4. Secondary Outcome: Number of Participants in Each Category of Clinical and Demographic Characteristics
Description: Clinical and demographic characteristics included gender, race, disease classification (relapsing remitting multiple sclerosis [RRMS], Secondary Progressive Multiple Sclerosis [SPMS], unknown & no MS disease), Prior use of DMDs & high-disease activity (HAD) status, education level and employment status. Number of participants in each category of clinical and demographic characteristics were reported in form of long term responders & non-responder. Here long term responder is defined as participants not requiring DMD 4 years or later following their last dose of IMP in parent study. Non-responder is defined as study participants requiring DMD < 4 years following their last dose of IMP in parent study.
Time Frame: as for outcome 3
Population: FAS included all participants participating in CLASSIC study [randomized in CLARITY and have received ≥ 1 course of IMP (Cladribine Tablets or placebo) or participants randomized in the ORACLE study and have received ≥ 1 course of IMP]. Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure and "Number analyzed" refers to number of participants evaluable for specified categories.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A
Number analyzed (Participants) | 627
Participants
  Long term responder: Sex (Female): number analyzed (Participants) | 378
  Long term responder: Sex (Female) | 251
  Non-responder: Sex (Female): number analyzed (Participants) | 249
  Non-responder: Sex (Female) | 171
  Long-term responder: Sex (Male): number analyzed (Participants) | 378
  Long-term responder: Sex (Male) | 127
  Non-responder: Sex (Male): number analyzed (Participants) | 249
  Non-responder: Sex (Male) | 78
  Long term responder: Race (White): number analyzed (Participants) | 378
  Long term responder: Race (White) | 368
  Non-responder: Race (White): number analyzed (Participants) | 249
  Non-responder: Race (White) | 244
  Long term responder: Race (Black or African American): number analyzed (Participants) | 378
  Long term responder: Race (Black or African American) | 1
  Non-responder: Race (Black or African American): number analyzed (Participants) | 249
  Non-responder: Race (Black or African American) | 0
  Long term responder: Race (Asian): number analyzed (Participants) | 378
  Long term responder: Race (Asian) | 5
  Non-responder: Race (Asian): number analyzed (Participants) | 249
  Non-responder: Race (Asian) | 3
  Long term responder: Race (Other): number analyzed (Participants) | 378
  Long term responder: Race (Other) | 4
  Non-responder: Race (Other): number analyzed (Participants) | 249
  Non-responder: Race (Other) | 2
  Long term responder: Type of MS-RRMS: number analyzed (Participants) | 378
  Long term responder: Type of MS-RRMS | 259
  Non-responder: Type of MS-RRMS: number analyzed (Participants) | 249
  Non-responder: Type of MS-RRMS | 173
  Long term responder: Type of MS-SPMS: number analyzed (Participants) | 378
  Long term responder: Type of MS-SPMS | 71
  Non-responder: Type of MS-SPMS: number analyzed (Participants) | 249
  Non-responder: Type of MS-SPMS | 41
  Long term responder: Type of MS-Unknown: number analyzed (Participants) | 378
  Long term responder: Type of MS-Unknown | 0
  Non-responder: Type of MS -Unknown: number analyzed (Participants) | 249
  Non-responder: Type of MS -Unknown | 14
  Long term responder: Type of MS-No MS disease: number analyzed (Participants) | 378
  Long term responder: Type of MS-No MS disease | 48
  Non-responder: Type of MS-No MS disease: number analyzed (Participants) | 249
  Non-responder: Type of MS-No MS disease | 21
  Long term responder: Prior Use of DMDs: number analyzed (Participants) | 276
  Long term responder: Prior Use of DMDs | 57
  Non-responder: Prior Use of DMDs: number analyzed (Participants) | 132
  Non-responder: Prior Use of DMDs | 33
  Long term responder: HDA participants: number analyzed (Participants) | 276
  Long term responder: HDA participants | 83
  Non-responder: HDA participants: number analyzed (Participants) | 132
  Non-responder: HDA participants | 35
  Long term responder: Education level (Below 8 Years): number analyzed (Participants) | 373
  Long term responder: Education level (Below 8 Years) | 19
  Non-responder: Education level (Below 8 Years): number analyzed (Participants) | 245
  Non-responder: Education level (Below 8 Years) | 16
  Long term responder: Education level (8 to 10 Years): number analyzed (Participants) | 373
  Long term responder: Education level (8 to 10 Years) | 73
  Non- responder: Education level (8 to 10 Years): number analyzed (Participants) | 245
  Non- responder: Education level (8 to 10 Years) | 43
  Long term responder: Education level (10 to 15 Years): number analyzed (Participants) | 373
  Long term responder: Education level (10 to 15 Years) | 190
  Non-responder: Education level (10 to 15 Years): number analyzed (Participants) | 245
  Non-responder: Education level (10 to 15 Years) | 130
  Long term responder: Education level (Over 15 Years): number analyzed (Participants) | 373
  Long term responder: Education level (Over 15 Years) | 91
  Non-responder: Education level (Over 15 Years): number analyzed (Participants) | 245
  Non-responder: Education level (Over 15 Years) | 56
  Long term responder: Employment Status (Employed for wages): number analyzed (Participants) | 378
  Long term responder: Employment Status (Employed for wages) | 160
  Non-responder: Employment Status (Employed for wages): number analyzed (Participants) | 249
  Non-responder: Employment Status (Employed for wages) | 122
  Long term responder: Employment Status (Self-Employed): number analyzed (Participants) | 378
  Long term responder: Employment Status (Self-Employed) | 38
  Non-responder: Employment Status (Self-Employed): number analyzed (Participants) | 249
  Non-responder: Employment Status (Self-Employed) | 17
  Long term responder: Employment Status (Out of Work for more than 1 year): number analyzed (Participants) | 378
  Long term responder: Employment Status (Out of Work for more than 1 year) | 12
  Non-responder: Employment Status (Out of Work for more than 1 year): number analyzed (Participants) | 249
  Non-responder: Employment Status (Out of Work for more than 1 year) | 13
  Long term responder: Employment Status (Out of Work for less than 1 year): number analyzed (Participants) | 378
  Long term responder: Employment Status (Out of Work for less than 1 year) | 4
  Non-responder: Employment Status (Out of Work for less than 1 year): number analyzed (Participants) | 249
  Non-responder: Employment Status (Out of Work for less than 1 year) | 2
  Long term responder: Employment Status (A Homemaker): number analyzed (Participants) | 378
  Long term responder: Employment Status (A Homemaker) | 22
  Non-responder: Employment Status (A Homemaker): number analyzed (Participants) | 249
  Non-responder: Employment Status (A Homemaker) | 24
  Long term responder: Employment Status (Retired): number analyzed (Participants) | 378
  Long term responder: Employment Status (Retired) | 67
  Non-responder: Employment Status (Retired): number analyzed (Participants) | 249
  Non-responder: Employment Status (Retired) | 19
  Long term responder: Employment Status (Unable to work): number analyzed (Participants) | 378
  Long term responder: Employment Status (Unable to work) | 48
  Non-responder: Employment Status (Unable to work): number analyzed (Participants) | 249
  Non-responder: Employment Status (Unable to work) | 26
  Long term responder: Employment Status (Not collected at the site): number analyzed (Participants) | 378
  Long term responder: Employment Status (Not collected at the site) | 3
  Non-responder: Employment Status (Not collected at the site): number analyzed (Participants) | 249
  Non-responder: Employment Status (Not collected at the site) | 6
  Long term responder: Employment Status (Unknown/Not reported): number analyzed (Participants) | 378
  Long term responder: Employment Status (Unknown/Not reported) | 24
  Non-responder: Employment Status (Unknown/Not reported): number analyzed (Participants) | 249
  Non-responder: Employment Status (Unknown/Not reported) | 20

5. Secondary Outcome: Clinical Characteristic: Expanded Disability Status Scale (EDSS) Score
Description: EDSS is a scale based on standardized neurological examination which comprised of optic, brain stem, pyramidal, cerebellar, sensory & cerebral functions, as well as walking ability. EDSS scores range from 0.0 (normal) to 10.0 (dead). Clinical characteristics of EDSS score in form of long-term responders & non-responder was reported for at parent study baseline (based on retrospective data collection [based on chart review] at study visit 1) & study visit 1. Here long term responder is defined as study participants not requiring DMD 4 years or later following their last dose of IMP in parent study. Non-responder is defined as study participants requiring DMD < 4 years following their last dose of IMP in parent study.
Time Frame: as for outcome 3
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cohort A
Number analyzed (Participants) | 627
score on a scale
  Long-term responders: EDSS score at parent study baseline: number analyzed (Participants) | 378
  Long-term responders: EDSS score at parent study baseline | 2.44 (1.292)
  Non-responders: EDSS score at parent study baseline: number analyzed (Participants) | 249
  Non-responders: EDSS score at parent study baseline | 2.38 (1.251)
  Long term responder: EDSS score at study visit 1: number analyzed (Participants) | 366
  Long term responder: EDSS score at study visit 1 | 3.23 (2.121)
  Non-responder: EDSS score at study visit 1: number analyzed (Participants) | 234
  Non-responder: EDSS score at study visit 1 | 3.32 (2.102)

6. Secondary Outcome: Clinical Characteristic: Number of Relapses
Description: Relapse was defined as participant-reported symptoms & objectively observed signs typical of an acute inflammatory demyelinating event in CNS, developing acutely or sub-acutely with duration of at least 24 hours, in absence of fever or infection. Clinical characteristics of number of relapses during last year before enrollment of parent study (it is reported based on retrospective data collection [based on chart review] at study visit 1) in the form of long-term responders & non-responder was reported. Here long term responder is defined as study participants not requiring DMD 4 years or later following their last dose of IMP in parent study. Non-responder is defined as study participants requiring DMD less than 4 years following their last dose of IMP in parent study.
Time Frame: as for outcome 3
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Relapses
Arm/Group | Cohort A
Number analyzed (Participants) | 408
Relapses
  Long-term responders: number of relapses during last year before enrollment of parent study: number analyzed (Participants) | 276
  Long-term responders: number of relapses during last year before enrollment of parent study | 1.3 (0.64)
  Non-responders: number of relapses during last year before enrollment of parent study: number analyzed (Participants) | 132
  Non-responders: number of relapses during last year before enrollment of parent study | 1.3 (0.56)

7. Secondary Outcome: Number of Total T1-weighted (T1-W) Lesions
Description: Total number of T1-W lesion were measured by Using magnetic resonance imaging (MRI) Scans. Here long term responder is defined as study participants not requiring DMD 4 years or later following their last dose of IMP in parent study. Non-responder is defined as study participants requiring DMD less than 4 years following their last dose of IMP in parent study.
Time Frame: At study visit 2, within 6 months from screening (Retrospective analysis of medical record of parent study-NCT00213135, NCT00641537 and NCT00725985)
Population: The MRI analysis population includes all FAS participants who signed the MRI sub- study informed consent. Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure and "Number analyzed" refers to number of participants evaluable for specified categories.
Measure: Mean (Standard Deviation); unit: lesions
Arm/Group | Cohort A
Number analyzed (Participants) | 39
lesions
  Long-term responder: number analyzed (Participants) | 20
  Long-term responder | 12.7 (8.97)
  Non-responder: number analyzed (Participants) | 19
  Non-responder | 16.1 (10.90)

8. Secondary Outcome: Number of Total T2-weighted (T2-W) Lesions
Description: Total number of T2-W lesion were measured by Using magnetic resonance imaging (MRI) Scans. Here long term responder is defined as study participants not requiring DMD 4 years or later following their last dose of IMP in parent study. Non-responder is defined as study participants requiring DMD less than 4 years following their last dose of IMP in parent study.
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: lesions
Arm/Group | Cohort A
Number analyzed (Participants) | 41
lesions
  Long-term responder: number analyzed (Participants) | 22
  Long-term responder | 20.2 (18.67)
  Non-responder: number analyzed (Participants) | 19
  Non-responder | 25.1 (18.17)

9. Secondary Outcome: T1-weighted (T1-W) Lesion Volume
Description: T1-W lesion volume were measured by Using magnetic resonance imaging (MRI) Scans. Here long term responder is defined as study participants not requiring DMD 4 years or later following their last dose of IMP in parent study. Non-responder is defined as study participants requiring DMD less than 4 years following their last dose of IMP in parent study.
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: cubic centimeter (cm^3)
Arm/Group | Cohort A
Number analyzed (Participants) | 38
cubic centimeter (cm^3)
  Long-term responder: number analyzed (Participants) | 20
  Long-term responder | 1.655 (1.3953)
  Non-responder: number analyzed (Participants) | 18
  Non-responder | 6.773 (6.4788)

10. Secondary Outcome: T2-weighted (T2-W) Lesion Volume
Description: T2-W lesion volume were measured by Using magnetic resonance imaging (MRI) Scans. Here long term responder is defined as study participants not requiring DMD 4 years or later following their last dose of IMP in parent study. Non-responder is defined as study participants requiring DMD less than 4 years following their last dose of IMP in parent study.
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: cubic centimeter (cm^3)
Arm/Group | Cohort A
Number analyzed (Participants) | 41
cubic centimeter (cm^3)
  Long-term responder: number analyzed (Participants) | 22
  Long-term responder | 4.920 (6.7665)
  Non-responder: number analyzed (Participants) | 19
  Non-responder | 14.664 (13.8109)

11. Secondary Outcome: Total Brain Volume
Description: Brain volume were measured by Using magnetic resonance imaging (MRI) Scans. Here long term responder is defined as study participants not requiring DMD 4 years or later following their last dose of IMP in parent study. Non-responder is defined as study participants requiring DMD less than 4 years following their last dose of IMP in parent study.
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: cubic centimeter (cm^3)
Arm/Group | Cohort A
Number analyzed (Participants) | 39
cubic centimeter (cm^3)
  Long-term responder: number analyzed (Participants) | 21
  Long-term responder | 1472.559 (59.9500)
  Non-responder: number analyzed (Participants) | 18
  Non-responder | 1417.431 (109.8668)

ADVERSE EVENTS:
Time Frame: Up to study visit 2 (Up to approximately 6 months and Retrospective AEs data collection based on chart review of participants from end of parent studies; NCT00213135, NCT00641537 and NCT00725985)
Arm/Group | Cohort A
All-Cause Mortality (participants affected / at risk) | 0/662
Serious Adverse Events (participants affected / at risk) | 1/662
Other Adverse Events (participants affected / at risk) | 8/662
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A (N=662)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A (N=662)
Lymphopenia (Blood and lymphatic system disorders) | 2
Leukopenia (Blood and lymphatic system disorders) | 2
Neutropenia (Blood and lymphatic system disorders) | 1
Nasopharyngitis (Infections and infestations) | 1
Autoimmune thyroid disorder (Endocrine disorders) | 1
Hepatic enzyme increased (Investigations) | 1
Flushing (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-07-03): https://cdn.clinicaltrials.gov/large-docs/04/NCT03961204/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-10): https://cdn.clinicaltrials.gov/large-docs/04/NCT03961204/SAP_001.pdf